CLINICAL TRIAL: NCT02032550
Title: Treatment Preference and Patient Centered Prostate Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCC201
Record Dates: First submitted 2013-12-23; First posted 2014-01-10 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Localized prostate cancer; Patient preference; Treatment choice; Decision making; Patient centered outcomes
MeSH Terms: conditions — Prostatic Neoplasms; Patient Preference

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preference Based Decision Aid (Experimental): The experimental arm of preference based decision aid intervention will complete a web-based conjoint analysis instrument for preference assessment.
  Interventions: Other: Preference Based Decision Aid
- Usual Care (No Intervention): Participants randomized into this group will have usual care from their doctors without any intervention

INTERVENTIONS:
Other: Preference Based Decision Aid — The objective of the preference based decision aid is to assess the treatment preferences of prostate cancer patients. The investigators will analyze the association between preferences, treatment choice and objective and subjective outcomes. The preference based decision aid will lead to a values-based patient centered treatment decision making. This will ultimately improve clinical decision making, clinical policy process, enhance patient centered care and improve prostate cancer outcomes.
  Arms: Preference Based Decision Aid

SUMMARY:
The purpose of this study is to develop a preference based decision aid to assess the treatment preferences of prostate cancer patients, and to analyze the interaction of treatment preferences, type of treatment received and their relationship with health related quality of life, satisfaction with care, decision regret, and psychological health of men with localized prostate cancer.

DETAILED DESCRIPTION:
The objective is to test the comparative effectiveness of a conjoint analysis decision aid intervention compared to usual care. The investigators will identify preferred attributes of prostate cancer treatments that will help in designing a conjoint analysis decision aid to help patients weigh treatment attributes. The investigators will employ values markers to represent clusters of values for particular aspects of treatments that are valued most by individual patients. The investigators will test if the concordance between values markers and treatment received is predictive of objective outcomes and subjective outcomes. The study hypothesis is that conjoint task may help in treatment choice and prostate cancer patients whose treatment is more concordant with their values markers will have improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with non-metastatic prostate cancer
2. Has not yet started radiation or surgery
3. Provide informed consent

Exclusion Criteria:

1. Distant, metastatic prostate cancer at diagnosis
2. Has already begun treatment for prostate cancer
3. Unable to communicate in English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2013-06; Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravishankar Jayadevappa, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Philadelphia Veteran's Affairs Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Chhatre S, Jefferson A, Cook R, Meeker CR, Kim JH, Hartz KM, Wong YN, Caruso A, Newman DK, Morales KH, Jayadevappa R. Patient-centered recruitment and retention for a randomized controlled study. Trials. 2018 Mar 27;19(1):205. doi: 10.1186/s13063-018-2578-7. PMID 29587805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preference Based Decision Aid | Usual Care
Started | 371 | 372
Completed | 343 | 350
Not Completed | 28 | 22

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes all participants that were randomized to the intervention group or to the usual care group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Preference Based Decision Aid | Usual Care | Total
Number analyzed (Participants) | 371 | 372 | 743
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.0) | 63.5 (7.6) | 63.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 371 | 372 | 743
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 355 | 351 | 706
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 51 | 102
  White | 306 | 295 | 601
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 371 | 372 | 743
Satisfaction with care [Mean (Standard Deviation); unit: units on a scale] — In the Patient Satisfaction Questionnaire (PSQ-18) survey, 18 items are consolidated into seven subscales to assess satisfaction with medical care and six aspects of care. The subscale score ranges between 1 and 5, with a higher score indicating higher satisfaction. The PSQ-18 has demonstrated good internal consistency (Cronbach's a, .86) and excellent test-retest reliability (r, 0.92).
  units on a scale | 3.96 (0.74) | 3.80 (0.81) | 3.88 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in Satisfaction With Care
Description: The investigators will measure Satisfaction with Care (PSQ-18). : The PSQ-18 scale measures satisfaction with care at baseline 3, 6, 12, and 24 months. Higher score indicates better satisfaction with care. Positive change indicates improvement in satisfaction with care.
Time Frame: baseline, 3, 6, 12 and 24 months
Population: All participants from both groups who were analyzed at end of 24 month follow-up.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Preference Based Decision Aid | Usual Care
Number analyzed (Participants) | 343 | 350
units on a scale
  Change at 3 month | 0.26 (0.05) | 0.07 (0.05)
  Change at 6 month | 0.28 (0.05) | 0.06 (0.05)
  Change at 12 month | 0.31 (0.05) | 0.15 (0.05)
  Change at 24 month | 0.44 (0.06) | 0.07 (0.06)

2. Secondary Outcome: Generic Health Related Quality of Life (HRQoL)
Description: Generic HRQoL data is obtained from Medical Outcome Study Short Form (SF-36) that assesses 8 health domains. Scores on each domain range from 0 to 100, higher scores indicating better generic HRQoL. Change in SF-36 domain scores between baseline to 24 month will be calculated as score at 24 month-score minus score at baseline. Positive change value indicates improvement in HRQoL from baseline to 24 month.
Time Frame: baseline to 24 month
Population: All participants from both groups were analyzed at 24 month. Change in scores on domain of Physical Function is reported below.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preference Based Decision Aid | Usual Care
Number analyzed (Participants) | 343 | 350
score on a scale | -0.13 (1.4) | -2.9 (1.3)

3. Secondary Outcome: Anxiety
Description: Anxiety will be measured using Memorial Anxiety Scale for Prostate Cancer (MAX-PC) scale
Time Frame: baseline, 3, 6, 12, and 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Urinary Symptoms
Description: The American Urological Association Symptom Index (AUA-SI) will be used to measured urinary symptoms
Time Frame: baseline, 3, 6, 12, and 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Treatment Choice
Description: The investigators will obtain data on primary and secondary treatments received, such as active surveillance, radical prostatectomy (RP), robotic-assisted laparoscopic prostatectomy (RALP), external beam radiation therapy (EBRT), brachytherapy (BT) or proton therapy (PT) via self report and verified from medical chart review.
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Depression
Description: The Center for Epidemiologic Studies Depression (CES-D) scale will be used to measure depression.
Time Frame: baseline, 3, 6, 12, and 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Satisfaction With Decision
Description: The Satisfaction with Decision (SWD) will be used to measure satisfaction with decision at 3, 6, 12 and 24 months.
Time Frame: baseline, 3, 6, 12, and 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Prostate Specific Health Related Quality of Life (HRQoL)
Description: Prostate specific HRQoL data is obtained from Expanded Prostate Cancer Index (EPIC), and measures four broad domains of urinary, bowel, sexual and hormonal symptoms. Scores on each sub-scale range from 0 to 100, with higher scores indicating better prostate cancer HRQoL. Proportion of participants returning to baseline scores will be calculated by comparing scores at baseline and at 24 month. Higher proportion indicates higher number of participants recovering baseline function by 24 month.
Time Frame: Baseline to 24 month
Population: All participants from both groups were analyzed at 24 month. Proportion returning to baseline scores is reported for domain of urinary function below.
Measure: Number; unit: Proportion of participants
Arm/Group | Preference Based Decision Aid | Usual Care
Number analyzed (Participants) | 343 | 350
Proportion of participants | 59.4 | 50

9. Other Pre Specified Outcome: Preference for Participation in Treatment Decision
Description: The Control Preferences Scale (CPS) assesses the role that patients want to play and perceive playing in treatment decisions.
Time Frame: baseline, 3, 6, 12, and 24 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Decision Conflict
Description: The Decision Conflict Scale (DCS) will be used to measure decision conflict.
Time Frame: 12 and 24 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Physician Trust
Description: The Patient Trust-Wake Forest Physician Trust Scale will be used to measure trust
Time Frame: baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Preference Based Decision Aid | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/371 | 4/372
Serious Adverse Events (participants affected / at risk) | 0/371 | 0/372
Other Adverse Events (participants affected / at risk) | 0/371 | 0/372

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT02032550/Prot_SAP_000.pdf